CLINICAL TRIAL: NCT03257488
Title: Screening of Obstructive Sleep Apnea Syndrome in Patients With Resistant Systemic Arterial Hypertension: Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Francesco Tavalazzi, Medical Doctor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 163/2014/O/Disp
Record Dates: First submitted 2017-02-10; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-07

CONDITIONS: Sleep Apnea, Obstructive; Resistant Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Screening device-Traditional device (Active Comparator): The patients included in the A Group will be studied during the first night with the screening device (type IV portable monitoring Somnocheck micro Weinmann) and with the traditional one during the following night.
  Interventions: Device: type IV portable monitoring (Somnocheck micro Weinmann)
- Traditional device-Screening device (Active Comparator): The patients included in the B Group will be studied during the first night with the traditional device and with the screening one (type IV portable monitoring Somnocheck micro Weinmann) during the following night.
  Interventions: Device: type IV portable monitoring (Somnocheck micro Weinmann)

INTERVENTIONS:
Device: type IV portable monitoring (Somnocheck micro Weinmann) — Somnocheck micro Weinmann: a screening device for sleep disorders assessment. Somnocheck 2 Weinmann: a diagnostic device for obstructive sleep apnea.
  Other Names: type III portable monitoring (Somnocheck 2 Weinmann)

SUMMARY:
This study evaluates the utility and reliability of Somnocheck micro Weinmann for obstructive sleep apnea syndrome (OSAS) screening in patients affected by resistant systemic arterial hypertension. Results are compared with a modified portable sleep apnea testing (type III portable monitoring: Somnocheck 2 Weinmann).

DETAILED DESCRIPTION:
OSAS is a syndrome characterized by the partial or total collapse of the high airways which determines snore, airflow limitation, hypopnea and apnea.These events cause desaturations, daytime sleepiness and an increased risk of cardio and cerebral vascular diseases.

OSAS's prevalence is estimated between 64-83% among patients affected by resistant arterial hypertension; therefore OSAS's screening is mandatory during the clinical work-up of these patients.

This study is a randomized, interventional, spontaneous, exploratory, cross-over and monocentric trial, which assesses the utility and reliability of the reduced cardio-respiratory monitoring (type IV portable monitoring: Somnocheck micro Weinmann) to estimate the prevalence of OSAS among patients affected by resistant systemic arterial hypertension. The results are compared with a complete cardio-respiratory monitoring (type III portable monitoring: Somnocheck 2 Weinmann).

ELIGIBILITY:
Inclusion Criteria:

* Resistant Arterial Hypertension
* Patients must sign the informed consent

Exclusion Criteria: ,

* atrial fibrillation with haemodynamic instability
* congestive hearth failure,
* BMI>45 kg/m2,
* respiratory failure
* renal or liver failure,
* stroke,
* implantable cardioverter-defibrillator (ICD),
* pacemaker (PM),
* previous diagnosis of OSAS,
* pregnancy,
* breastfeeding,
* patients must not be already enrolled in other clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Apnea hypopnea index (AHI) differences between screening device and the traditional diagnostic one. | These two procedures must be done in the same patient within 5 days
  Apnea hypopnea index (AHI) differences between screening device and the traditional diagnostic one.

SECONDARY OUTCOMES:
Number of Participants with cardiovascular abnormalities 1 | Cardiovascular assessment must be done within 6 months before the sleep studies.
  Number of Participants with cardiovascular abnormalities assessed by arterial blood pressure monitoring
Number of Participants with cardiovascular abnormalities 2 | Cardiovascular assessment must be done within 6 months before the sleep studies.
  Number of Participants with cardiovascular abnormalities assessed by ecocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda ospedaliera policlinico Sant'Orsola-Malpighi, Bologna, Italy